CLINICAL TRIAL: NCT06040892
Title: Spatial Hearing Rehabilitation in Noise for Bilateral Cochlear Implant Children
Acronym: KidTrain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL22_0893
Record Dates: First submitted 2023-08-30; First posted 2023-09-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cochlear Implantation
Keywords: spatial hearing; virtual reality; hearing loss; rehabilitation
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): bilateral cochlear implant children with rehabilitation including 8 sessions with a spatialized sensory index
  Interventions: Diagnostic Test: SPHERE protocol : Spatial hearing performances test; Diagnostic Test: FRASIMAT Test : audiology test of speech in noise perception; Diagnostic Test: Kid SSQ questionnaire of life : The Speech, Spatial and Other Qualities of Hearing Scale; Other: spatial hearing rehabilitation program
- Group B (Experimental): bilateral cochlear implant children with rehabilitation including initially 4 sessions without spatialized sensory cue followed by 4 sessions with spatialized sensory cue
  Interventions: Diagnostic Test: SPHERE protocol : Spatial hearing performances test; Diagnostic Test: FRASIMAT Test : audiology test of speech in noise perception; Diagnostic Test: Kid SSQ questionnaire of life : The Speech, Spatial and Other Qualities of Hearing Scale; Other: spatial hearing rehabilitation program
- Normal hearing volunteers (Active Comparator): Children without known hearing loss
  Interventions: Diagnostic Test: SPHERE protocol : Spatial hearing performances test; Diagnostic Test: FRASIMAT Test : audiology test of speech in noise perception; Diagnostic Test: Kid SSQ questionnaire of life : The Speech, Spatial and Other Qualities of Hearing Scale

INTERVENTIONS:
Diagnostic Test: SPHERE protocol : Spatial hearing performances test — Participants will be instructed to localize a sound emitted in their environment using a virtual reality setup (SPHERE protocol).
Diagnostic Test: FRASIMAT Test : audiology test of speech in noise perception — Intelligibility threshold is the signal-to-noise ratio (in decibels) for which the subject can repeat 50% of the words heard in a dichotic listening.
Diagnostic Test: Kid SSQ questionnaire of life : The Speech, Spatial and Other Qualities of Hearing Scale — The SSQ questionnaire is a clinical subjective scale that allows evaluating of hearing performances in daily life. The questionnaire is divided into 3 main items (A: speech; B: spatial hearing; C: other qualities of hearing) comprising questions with rating scores out of ten.
Other: spatial hearing rehabilitation program — The tool makes it possible to propose rehabilitation programs adapted to the performance and expectations of each child. This program will manipulate both the ambient sound with varying background noise to simulate daily life environments (i.e. making auditory detection more or less complex), and also manipulate virtual immersive environment (i.e. giving more or less relevant visual cues related to real sound location).
  Arms: Group A; Group B

SUMMARY:
In recent decades, there was a great expansion for bilateral cochlear implantation (bCI) in children, leading to an improvement of their quality of life. However, spatial hearing skills of bCI children remain limited, even for children with the best speech understanding outcomes. Recent studies have brought new insights in spatial hearing by using virtual reality to record spatial hearing performance in 3D and the impact of active listening (i.e. free head exploration during sound emission): all bCI children showed spatial hearing difficulties related to front-back confusions and distance perception, which partly resulted from the reduction in auditory cues by the CI settings. However, bCI children notably improved under conditions of active listening, suggesting that interaction with environment could represent a rehabilitation entry strategy to help bCI users when faced with complex auditory scenes in daily life.

The ability to localize sounds in space (spatial hearing) and the ability to understand speech in noise are both auditory skills essential in daily interactions with our physical and social environment and, when deficient, limit the quality of life. However, there is no specific rehabilitation program devoted to spatial hearing which could help children face their daily difficulties in noisy environments. Even though technological advances are crucial to improve the restoration of hearing functions, these improvements are also highly dependent on rehabilitation strategies to train our auditory brain to face the restoration of binaural processing or to decode the impoverished spectral information delivered by the CI.

The investigators recently performed a pilot study in bCI adults who attended 8 training sessions of spatial hearing, involving a sensorial and interactive immersive environment (i.e. virtual reality with auditory and visual environment during an active listening task). All participants benefitted of the training, in terms of spatial hearing performance, speech understanding in noise, and quality of life. All early benefits were maintained 1 month after the end of training.

The investigators aim to propose a spatial hearing rehabilitation program (KidTrain) adapted to bCI children from 8 to 17 years old, based on their previous pilot study on bCI adults. Their tool makes it possible to propose rehabilitation programs adapted to the performance and expectations of each child. This program will manipulate both the ambient sound with varying background noise to simulate daily life environments (i.e. making auditory detection more or less complex), and also manipulate virtual immersive environment (i.e. giving more or less relevant visual cues related to real sound location). The KidTrain's effects will be measured with different auditory tests performed in noisy environments. The investigators will also include Normal Hearing (NH) children as age-matched control groups to perform the auditory tests in noise. These NH groups will also bring new insights of spatial hearing maturation in complex auditory environments. Based on our preliminary data in bCI adults, this 'KidTrain program' should improve spatial hearing skills of bCI children, speech comprehension in noise and quality of life in many daily situations.

Virtual reality (VR) has recently proven its effectiveness in rehabilitation in many domains and recent studies have shown that this technology has its place in the auditory evaluation and adaptation of spatial hearing. This VR approach takes advantage of the control of multisensory cues of our environment (audio and visual) during a spatial hearing task, and allows the subject to interact with his environment according to his hearing abilities and needs (i.e. active listening).

Based on their previous study conducted in bCI and NH children and on their spatial training study conducted with bCI adults, the investigators wish to respond to the growing need of spatial hearing rehabilitation for bCI children. To achieve this goal, the investigators will improve the spatial training program by adding different immersive environment in VR with various background noise to simulate daily life environments. This approach will also be a great opportunity to characterize the developmental stages of spatial hearing maturation in NH children. Thus, this project will propose new axes of speech therapy on the Orthophonie & Surdité platform, combining spatial hearing and speech understanding in noise. This innovative and adapted rehabilitation program will lead the speech therapist to propose more adapted and effective rehabilitations for the daily life of deaf children.

ELIGIBILITY:
Inclusion Criteria:

* Child aged between 7 and 17 years
* Normal vision (including correction),
* Able to understand the experimental instructions,
* Parents or guardians informed of the study and having signed the consent form,

Specific for NH:

* Normal tone audiometry (mean threshold ≤ 30 dB). Specific for bIC
* Minimum 2 years of binaural experience,
* Average speech recognition ≥ 80% with both cochlear implants

Exclusion Criteria:

* Bilateral vestibular areflexia,
* Attention deficit disorder,
* Known neurological or psychiatric disorders,
* Oculomotor disorders,
* Parents not affiliated to a social security scheme or beneficiaries of a similar scheme who sign the consent for the child's participation,
* Subject participating in other interventional research with an exclusion period still ongoing at inclusion.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2027-07-27 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate the very short-term effects of spatial rehabilitation on the auditory performance of bCI children. | Immediately after 4 training sessions - day 42
  The effect of spatial rehabilitation will be defined as any change in auditory performance (SPHERE value), between the initial assessment and after 4 training sessions.
To evaluate the very short-term effects of spatial rehabilitation on the auditory performance of bCI children. | Immediately after 4 training sessions - day 42
  The effect of spatial rehabilitation will be defined as any change in auditory performance (FRASIMAT value), between the initial assessment and after 4 training sessions.
To evaluate the very short-term effects of spatial rehabilitation on the auditory performance of bCI children. | Immediately after 4 training sessions - day 42
  The effect of spatial rehabilitation will be defined as any change in auditory performance (KID-SSQ score), between the initial assessment and after 4 training sessions.

SECONDARY OUTCOMES:
To evaluate the compliance of bCI children with the rehabilitation protocol | At the end of the study ( Visit 13 - day 98)
  Number of training sessions attended by bCI patients
To evaluate the impact of a spatialized sensory index in rehabilitation. | At the end of the study ( Visit 13 - day 98)
  Measures obtained at the E2 assessment (SPHERE value) between the group of bCI children in group A and those in group B.
To evaluate the impact of a spatialized sensory index in rehabilitation. | At the end of the study ( Visit 13 - day 98)
  Measures obtained at the E2 assessment (FRASIMAT value) between the group of bCI children in group A and those in group B.
To evaluate the impact of a spatialized sensory index in rehabilitation. | At the end of the study ( Visit 13 - day 98)
  Measures obtained at the E2 assessment (KID-SSQ score) between the group of bCI children in group A and those in group B.
To evaluate the effect in the very short/short and medium term of spatial hearing rehabilitation on the spatial sound localization performance of bIC children compared to NH children | At evaluation visits Day 0, 42, 77 and 98
  SPHERE confusion rates (front-back, up-down, near-far) for bCI children at E2, E3 and E4 and NH children at E0.
To evaluate the effect of very short-term, short-term and medium-term spatial hearing rehabilitation on the speech comprehension performance of bIC children compared to NH children. | At evaluation visits Day 0, 42, 77 and 98
  FRASIMAT noise intelligibility scores for bCI children in E2, E3 and E4 and those for NH children in E0.
To evaluate the effect of very short-term and short-term and medium-term spatial hearing rehabilitation on the quality of life performance of bIC children compared to NH children. | At evaluation visits Day 0, 42, 77 and 98
  KID-SSQ spatial hearing scores obtained by bCI children in E2, E3 and E4 and those obtained by NH children in E0.
To assess the absence of spontaneous changes in auditory performance. | At day 0 and 7
  SPHERE measure for the bCI and NH groups between the E0 and E1 assessments.
To assess the absence of spontaneous changes in auditory performance. | At day 0 and 7
  FRASIMAT measure for the bCI and NH groups between the E0 and E1 assessments.
To assess the absence of spontaneous changes in auditory performance. | At day 0 and 7
  KID SSQ measure for the bCI and NH groups between the E0 and E1 assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie Coudert, MD, Study Chair — Hospices Civils de Lyon
Locations (1):
- Service d'Oto-Rhino-Laryngologie et Chirurgie cervico-faciale Hôpital Edouard Herriot, Groupement Hospitalier Centre, Lyon, France

REFERENCES:
- [Background] Yuzefovsky AI, Lonardo RF, Michel RG. Spatial discrimination against background with different optical systems for collection of fluorescence in laser-excited atomic fluorescence spectrometry with a graphite tube electrothermal atomizer. Anal Chem. 1995 Jul 1;67(13):2246-55. doi: 10.1021/ac00109a052. PMID 8694251
- [Background] Valzolgher C, Gatel J, Bouzaid S, Grenouillet S, Todeschini M, Verdelet G, Salemme R, Gaveau V, Truy E, Farne A, Pavani F. Reaching to Sounds Improves Spatial Hearing in Bilateral Cochlear Implant Users. Ear Hear. 2023 Jan-Feb 01;44(1):189-198. doi: 10.1097/AUD.0000000000001267. Epub 2022 Aug 19. PMID 35982520
- [Background] Coudert A, Verdelet G, Reilly KT, Truy E, Gaveau V. Intensive Training of Spatial Hearing Promotes Auditory Abilities of Bilateral Cochlear Implant Adults: A Pilot Study. Ear Hear. 2023 Jan-Feb 01;44(1):61-76. doi: 10.1097/AUD.0000000000001256. Epub 2022 Aug 9. PMID 35943235